CLINICAL TRIAL: NCT00258193
Title: A Phase 2 Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study of the Pharmacodynamic Effects of Orally Administered 100ug and 1000ug QD MD-1100 Acetate on Gastrointestinal Transit in Patients With Constipation Predominant Irritable Bowel Syndrome (C-IBS)
Brief Title: Phase 2 Study of MD-1100 Acetate on Gastrointestinal Transit in Patients With C-IBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol MCP-103-005
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: C-IBS; IBS-C; Constipation-predominant Irritable Bowel Syndrome; Constipation Predominant Irritable Bowel Syndrome; Irritable Bowel Syndrome; IBS; Transit; Scintigraphy; Gastroenterology; Gastrointestinal; GC; MD-1100 Acetate; MD-1100; linaclotide; linaclotide acetate
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — linaclotide

INTERVENTIONS:
Drug: MD-1100 Acetate

SUMMARY:
* The primary objective of this trial is to compare the dose-ranging pharmacodynamic effects of orally administered placebo, and 100 and 1000 ug qd of MD-1100 Acetate on gastrointestinal transit in patients with C-IBS.
* The secondary objectives of this trial are:

  1. To compare the dose ranging pharmacodynamic effects of placebo, and 100 and 1000 ug MD-1100 Acetate once daily on time to first bowel movement after first drug intake.
  2. To describe and summarize the effects of placebo, and 100 and 1000 ug MD-1100 Acetate once daily on stool frequency, stool consistency, ease of passage and sensation of incomplete evacuation during the Treatment Period relative to Baseline.

DETAILED DESCRIPTION:
Using a double-blind, randomized, placebo-controlled, parallel group study design, the effects of placebo and two different doses of orally administered MD-1100 Acetate on gastric emptying, small bowel transit and total colonic transit will be compared and evaluated in patients with C-IBS.

After eligibility is confirmed, the patient will return for baseline measurement of colonic transit to ensure that the transit profile is not greater than the mean transit profile of healthy controls in order to avoid a ceiling effect. A patient must have a geometric center of ≤2.65 at 24 hours, or ≤3.0 at 24 hours and ≤3.9 at 48 hours in order to be randomized to a 5-day Treatment Period of study medication. Eligible patients will receive oral study medication for 5 days during which colonic transit will be measured.

Approximately 36 (n=36) patients will be randomized to one of three different treatment groups: placebo (n=12), 100 ug MD-1100 (n=12), or 1000 ug MD-1100 (n=12). All dosing of study medication will be supervised at the Mayo Clinic.

Patients will complete a daily Stool Diary to record bowel habits for 5 consecutive days during the Pretreatment Period and then for the 5 consecutive days of the Treatment PeriodPhysical examinations, vital signs, electrocardiograms, and clinical laboratory tests will be performed throughout the study and adverse events will be recorded for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient agrees to use a medically accepted, double-barrier form of contraception (e.g., IUD and condom) during participation;
* No evidence of pelvic floor dysfunction and the completion of a negative digital rectal exam prior to the first dose of study medication;
* Absence of an evacuation disorder as defined per protocol;
* Patients must meet ROME II Criteria for C-IBS;
* The patient's Baseline Colonic Transit Test must show a geometric center (GC) ≤ 2.65 at 24 hours, or ≤ 3.0 at 24 hours and ≤ 3.9 at 48 hours.

Exclusion Criteria:

* History of clinically-significant manifestations of any major system organ class;
* History of inflammatory bowel disease or gastric ulcers;
* Significant GI surgery within 6 months;
* Clinically-significant prolonged diarrhea within 60 days;
* Special dietary habit and/or an intense physical workout program within 4 weeks;
* Certain drug hypersensitivities
* History of alcoholism or drug addiction within 12 months;
* Receipt of an investigational drug during the study or within 30 days;
* Use of any prescription medication or OTC, non-prescription medications disallowed by the protocol within 7 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2006-01; Study Completion 2006-09

PRIMARY OUTCOMES:
(Safety) AEs to be collected beginning with patient's first administration of study medication through final study visit
Clinical chemistry, hematology, and urinalyses to be performed before and after the Treatment Period
Cardiac safety will be monitored by ECG recordings
(Efficacy) Primary endpoints for analysis of efficacy are the colonic geometric center (GC) at 24 hours and ascending colon t1/2 values.

SECONDARY OUTCOMES:
Secondary transit endpoints will be gastric emptying t1/2, colonic filling at 6 hours, colonic GC at additional time points including 48 hours, and time to first bowel movement after the first dose of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic Foundation
Locations (1):
- Mayo Clinic Foundation, Rochester, Minnesota, United States